CLINICAL TRIAL: NCT05584774
Title: Clinical Outcomes of Percutaneous Endoscopic Lumbar Discectomy Add by Annuloplasty and Nucleoplasty for Lumbar Disc Herniation: Randomized Controlled Trial
Brief Title: Percutaneous Endoscopic Lumbar Discectomy Add by Annuloplasty and Nucleoplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Jatupon Kongtharvonskul, principle investigator, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NO40/2565
Record Dates: First submitted 2022-10-06; First posted 2022-10-18 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PELD (Placebo Comparator)
  Interventions: Procedure: PELDAN
- PELD and annuloplasty and nucleoplasty (Active Comparator)
  Interventions: Procedure: PELDAN

INTERVENTIONS:
Procedure: PELDAN — percutaneous endoscopic lumbar dissectomy and annuloplasty and nucleoplasty

SUMMARY:
Recently, percutaneous endoscopic lumbar discectomy (PELD) is also commonly performed for lumbar disc herniation. Following discectomy, the relief of leg pain is common; however, the relief of back pain is less predictable. The association of back pain and lumbar disc herniation is still unclear. PELD and Annuloplasty (PELDA) can relieve back pain associated with disc herniation as well as leg pain through decompression and thermal ablation of annular defects in selected patients. Another problem that rapidly increasing go along with the growing number of microdiscectomies is directly proportional to the number of patients who undergo re-operations due to recurrences. The surgical treatment can be helpful in prevention of re-operations is nucleoplasty. Endoscopic discectomy for lumbosacral herniation supplemented with nucleoplasty can reduce the recurrence and reoperation rates.

ELIGIBILITY:
Inclusion Criteria:

* Primary single-level lumbosacral intervertebral disc herniation at the L4-L5 or L5- S1 level will perform surgical intervention of percutaneous endoscopic lumbar discectomy
* All patients present with sciatica and back pain that will not improve with conservative treatment for a minimum of 6 weeks
* All patients undergo plain radiographs, magnetic resonance imaging (MRI)
* The patients will require to have an obvious disc herniation that caused compression of a nerve root corresponding to the dermatomal distribution of the leg symptoms.

Exclusion Criteria:

* Patients have foraminal, extra-disc herniation, multilevel disc herniation, spinal stenosis, spondylolisthesis, scoliosis, prior lumbar surgery, spinal infection, spinal tumor, and a history of hip or knee arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
VAS back pain | 48 weeks
VAS leg pain | 48 weeks

SECONDARY OUTCOMES:
ODI | 48 weeks
  Oswestry disability index
complications | 48 weeks
  Nerve injury, foot drop, dura tear
re-operation | 48 weeks

IPD SHARING:
Plan to Share IPD: No